CLINICAL TRIAL: NCT07371858
Title: The Effect of Home-Based Exercise on Sarcopenia Risk, Functional Capacity, Depression, Fatigue, Sleep, and Quality of Life in Chronic Kidney Disease Patients
Brief Title: The Effect of Home-Based Exercise on Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gokce Yagmur Gunes Gencer, Associate Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: The Effect of Exercise on CKD
Record Dates: First submitted 2025-04-22; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease Stage 4 and 5; Exercise; Home Based Care; Sarcopenia; Telehealth
Keywords: Chronic Kidney Disease stage 4 and 5; Home-Based Exercise; Functional Capacity; Sarcopenia; Telehealth
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Sarcopenia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Based Exercise Group (Experimental): Patients participating in the home-based exercise program
  Interventions: Other: Treatment
- Control Group (No Intervention): Patients not participating in the home exercise program

INTERVENTIONS:
Other: Treatment — The study group will be provided with a 12-week home exercise program. Participants will receive a home-based exercise program for 30-55 minutes per day, 3-4 times a week for 12 weeks, with the intensity of exercise adjusted based on the participant's perceived exertion. The program consists of warm-up and cool-down exercises, strength exercises (upper-lower extremities, abdominal-back muscles), and aerobic exercise. A website will be designed where patients can access and track their home exercise programs using predefined usernames and passwords. Patients will be able to watch exercise videos on the website. Additionally, patients will evaluate the difficulty of their daily exercises through their profiles on the website. For patients who cannot adhere to tracking via the website, exercise videos will be shared via the WhatsApp application. Exercise tracking will be done through the exercise schedule provided to patients.
  Arms: Home Based Exercise Group

SUMMARY:
The aim of this study is to investigate the effects of home-based exercise on the risk of sarcopenia, functional capacity, anxiety, depression, fatigue, sleep, and quality of life in patients aged 45 and over with chronic kidney disease (Stage 4-5) who are not on dialysis.

A total of 26 voluntary participants aged 45 and above with chronic kidney disease (Stages 4-5) who are not undergoing dialysis will be included in the study. Participants will be randomly assigned to either the intervention or control group using block randomization method. While the intervention group will engage in a 12-week home exercise program, the control group will not receive any exercise intervention. The effects of the 12-week home exercise program on Sarcopenia Risk, Functional Capacity, Depression, Fatigue, Sleep, and Quality of Life will be evaluated before and after the intervention in this study.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of home-based exercise on sarcopenia risk, functional capacity, anxiety, depression, fatigue, sleep, and quality of life in patients aged 45 and over with chronic kidney disease (Stage 4-5) who are not undergoing dialysis.

A total of 26 patients aged 45 and over with chronic kidney disease (Stage 4-5) who are not on dialysis and followed up at the Nephrology Outpatient Clinic, Low Clearance Department of Akdeniz University Hospital, will be included in the study as voluntary participants. The study and control groups will be determined using block randomization method.

Both groups will undergo SARC-F questionnaire, anthropometric measurements, Mini Nutritional Assessment Short Form (MNA-SF), FACIT fatigue scale, Hospital Anxiety and Depression Scale, Pittsburgh Sleep Quality Index, Kidney Disease Quality of Life Scale (KDQOL-SF), 6-minute walk test, 10-meter walk speed test, 5-repetition sit-to-stand test, handgrip strength measurement, and manual muscle strength measurements before the study (week 0). In addition to these assessments, the study group will receive a home-based exercise program for 30-55 minutes, 3-4 times a week for 12 weeks, with the intensity of exercise adjusted according to the participant's perceived exertion, and each participant will be supervised by a physiotherapist until they learn the exercises. After 12 weeks, all these questionnaires and tests will be repeated for both groups, and the results will be compared.

Additionally, in this study, a website will be designed to facilitate access to and monitoring of home-based exercise programs, enabling participants to benefit from telehealth services-a prominent topic in recent healthcare research. At the end of the intervention, the Exercise Adherence Rating Scale (EARS) will be administered to the intervention group to evaluate patients' adherence to the prescribed home exercise program, as well as the reasons for adherence or non-adherence. Through this assessment, the effectiveness of the implemented telehealth service will be measured. Therefore, this study emphasizes a personalized and comprehensive approach that not only addresses health-related outcomes but also aims to improve patients' overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being followed up at the Nephrology Outpatient Clinic, Low Clearance Department of Akdeniz University Hospital
* Being aged 45 and above
* Complying with the test protocols
* Obtaining a score of 24 or above on the MMSE for individuals aged 65 and above.

Exclusion Criteria:

* Individuals under the age of 45
* Those who have had coronary artery disease or stroke (CVA) in the last three months
* Individuals with chronic heart failure (Stage 3-4)
* Those with any neurological or orthopedic disease affecting independent walking ability
* Individuals aged 65 and over who score below 24 on the Mini Mental State Examination
* Those unable to comply with the test protocols.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | 0. week
  Individuals scoring 24 points or higher on the scale will be included in the study. The Mini-Mental State Examination (MMSE) is a widely used cognitive screening instrument with a minimum score of 0 and a maximum score of 30. Higher MMSE scores indicate better global cognitive functioning, reflecting more intact orientation, attention, memory, language, and visuospatial abilities. Conversely, lower scores are associated with greater cognitive impairment. The MMSE is commonly employed in both clinical practice and research to assess cognitive status and to monitor changes in cognitive performance over time.
Modified Borg Scale | 12 week
  Participants included in the study group will be instructed to rate the perceived intensity of their pre-exercise activities using the modified Borg Scale before starting the exercise program. They will be taught to record their ratings on the chart within their profile accounts on the specially designed website for the study, or if they cannot adapt to the website, they will be instructed to note them on the chart provided to them after each exercise session. The Modified Borg Scale is a subjective rating scale used to quantify perceived exertion or dyspnea during physical activity. The scale ranges from a minimum value of 0, indicating no perceived exertion or breathlessness, to a maximum value of 10, representing maximal or very severe exertion or dyspnea. Higher scores on the Modified Borg Scale reflect greater symptom severity and therefore indicate a worse perceived physiological response to activity.
SARC-F Questionnaire | 0.-12. week
  The SARC-F, a screening test for sarcopenia, will be administered to both the study and control groups before and after the program. The SARC-F Questionnaire is a brief, self-reported screening tool used to identify individuals at risk of sarcopenia. The total score ranges from a minimum of 0 to a maximum of 10, based on five items assessing strength, assistance with walking, rising from a chair, stair climbing, and falls. Higher SARC-F scores indicate poorer muscle function and a greater likelihood of sarcopenia, whereas lower scores reflect better physical performance. A total score of 4 or higher is commonly used as a cutoff to suggest an increased risk of sarcopenia.
Anthropometric Measurement | 0.-12. week
  Anthropometric assessments will be conducted as separate outcome measures, each reported with its corresponding unit of measurement. Body weight (kg) and height (m) will be measured independently and will be used to calculate body mass index (BMI, kg/m²) as a derived outcome. In addition, waist circumference (cm), upper arm circumference (cm), and calf circumference (cm) will be assessed as distinct measures of body composition and muscle mass. Each anthropometric variable will be evaluated individually to assess changes in the participant's health status and physical condition before and after the program.
Mini Nutritional Assessment-Short Form (MNA-SF) | 0.- 12. week
  The Mini Nutritional Assessment-Short Form (MNA-SF) is a validated screening tool used to evaluate nutritional status in older adults. The total score ranges from a minimum of 0 to a maximum of 14. Higher MNA-SF scores indicate better nutritional status, reflecting adequate intake, stable weight, preserved mobility, and absence of psychological stress or acute disease. In contrast, lower scores are associated with malnutrition or risk of malnutrition. Commonly used thresholds classify scores of 12-14 as normal nutritional status, 8-11 as at risk of malnutrition, and 0-7 as malnourished. This questionnaire will be administered to both groups before and after the study, and the results will be compared.
The Kidney Disease Quality of Life Short Form (KDQOL-SF) | 0.- 12. week
  The KDQOL-SF consists of 80 items divided into 19 dimensions. Scores in each dimension range from 0 to 100, with higher scores reflecting better quality of life. This questionnaire will be administered to both groups before and after the study, and the results will be compared.
Hospital Anxiety and Depression Scale (HADS) | 0.- 12. week
  The Hospital Anxiety and Depression Scale (HADS) is a self-administered instrument designed to assess symptoms of anxiety and depression in clinical populations. It consists of 14 items, divided into two subscales: HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D), each comprising seven items. Scores for each subscale range from a minimum of 0 to a maximum of 21, yielding a possible total score range of 0 to 42. Higher scores indicate greater severity of anxiety and depressive symptoms and therefore represent a worse psychological outcome, whereas lower scores reflect fewer symptoms and better emotional well-being. The questionnaire will be administered to both groups before and after the study for comparison.
FACIT Fatigue Scale | 0.- 12. week
  The FACIT Fatigue Subscale is a 13-item scale that measures the level of fatigue experienced by an individual during their daily activities over the past seven days. Fatigue level is measured on a four-point Likert scale (4 = Not at all tired, 0 = Very tired). The score range is 0-52, with a score of less than 30 indicating severe fatigue. The higher the score, the better the quality of life. The scale will be administered to both groups before and after the study, and the results will be compared.
Pittsburgh Sleep Quality Index (PSQI) | 0.- 12. week
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized self-report instrument used to assess sleep quality and sleep disturbances over the previous month. The PSQI yields a global score ranging from a minimum of 0 to a maximum of 21, derived from seven component scores. Higher PSQI scores indicate poorer sleep quality and more severe sleep disturbances, whereas lower scores reflect better overall sleep quality. A global PSQI score greater than 5 is commonly used to distinguish poor sleepers from good sleepers in both clinical and research settings. The scale will be administered to both groups before and after the study, and the results will be compared.
6-Minute Walk Test | 0.- 12. week
  The 6-Minute Walk Test measures the distance a patient can walk quickly within a 6-minute period. It is conducted in a straight corridor of at least 30 meters, where the patient walks as quickly as possible without running. The distance walked is measured. Additionally, oxygen saturation and pulse will be monitored using a pulse oximeter before exercise, after exercise, and as needed during exercise. The test will be conducted before and after the study for both groups.
10-Meter Walk Test | 0.-12. week
  10-Meter Walk Test is used to assess an individual's physical capacity. The test measures the time it takes for the person to walk a distance of 10 meters. The individual is asked to walk the 10 meters at their own normal pace and return to the starting line as quickly as possible. The measurement is repeated twice, and the best result is recorded and interpreted. The test will be conducted before and after the study for both groups, and the results will be compared.
Five Times Sit to Stand Test | 0.- 12. week
  In this test, a standard chair is used to determine the speed of sitting and standing. Participants are asked to "stand up and sit down 5 times as quickly as possible." The time from the start of the movement to the completion of the 5th standing position is measured in seconds using a stopwatch. Two repetitions are performed, and the average of these 2 values is taken. This test is conducted to assess participants' lower extremity muscle strength and mobility, providing information about their functional capacity. The test will be conducted before and after the study for both groups, and the results will be compared.
Manual Muscle Testing | 0.- 12. week
  Manual Muscle Testing (MMT) is a clinical assessment method used to evaluate voluntary muscle strength. Muscle strength is typically graded on an ordinal scale ranging from a minimum score of 0 to a maximum score of 5. A score of 0 indicates no visible or palpable muscle contraction, while a score of 5 represents normal muscle strength against full resistance. Higher MMT scores reflect greater muscle strength and better functional performance, whereas lower scores indicate varying degrees of muscle weakness. MMT is widely used in clinical practice and research to assess neuromuscular function and to monitor changes in muscle strength over time. Patients included in the study will be evaluated for muscle strength in shoulder flexors/extensors, elbow flexors/extensors, wrist flexors/extensors, hip flexors/extensors, knee flexors/extensors, and ankle dorsiflexors/plantar flexors. Both groups will be assessed before and after the study, and the results will be compared.
Hand Grip Strength | 0.- 12. week
  This measurement, to be conducted on both groups, will interpret hand grip strength obtained with a hand dynamometer based on these cutoff points, and values before and after the study will be compared.
Blood parameters | 0.- 12. week
  At the beginning and end of the study, routine laboratory parameters will be evaluated as separate outcome measures, each reported using its standard unit of measurement. These will include complete blood count parameters (reported individually according to standard hematological units), serum calcium (mg/dL), serum phosphorus (mg/dL), parathyroid hormone (pg/mL), and serum creatinine (mg/dL). Each laboratory variable will be analyzed independently to assess changes in the patient's biochemical status over the course of the study, based on data obtained from the medical records.

SECONDARY OUTCOMES:
Exercise Adherence Rating Scale (EARS) | 12. week
  At the end of the 12-week period, the Exercise Adherence Rating Scale (EARS), developed by Newman-Beinart et al., will be applied to evaluate adherence to the home-based exercise program in the intervention group. The scale, designed for patients with chronic diseases, assesses adherence as well as reasons for adherence or non-adherence. It consists of three sections: Section A (6 unscored, customizable items), Section B (6 fixed items scored on a 5-point Likert scale; items 1, 4, and 6 reverse-scored; total score 0-24), and Section C (10 fixed items assessing barriers/supports for adherence; items 4, 5, 6, 7 reverse-scored; total score 0-40). The final adherence score is calculated by summing Sections B and C (range: 0-64), with higher scores indicating greater adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Gökçe Yağmur Güneş Gencer, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided